CLINICAL TRIAL: NCT00771706
Title: Longitudinal Study of Children With a Chronic Cough and the Impact of Gastroesophageal Reflux
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was not activated, no data was collected.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 04-12-076
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Cough; Gastroesophageal Reflux
Keywords: Pediatric Cough, Quality of Life; Drug (including placebo)
MeSH Terms: conditions — Cough; Gastroesophageal Reflux | interventions — Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proton Pump Inhibitor (Experimental): To compare the cough reduction rate using either PPI or placebo in children with a chronic cough.
  Interventions: Drug: Proton Pump Inhibitor
- Sugar Pill (Placebo Comparator): To compare the cough reduction rate using either PPI or placebo in children with a chronic cough
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proton Pump Inhibitor — The PPI arm will consist of a two week course of PPI at a dose 1mg/kg/dose twice daily (minimum dose: 7.5 mg BID; maximum dose: 30 mg BID)
  Other Names: PPI
  Arms: Proton Pump Inhibitor
Drug: Placebo — To compare the cough reduction rate using either PPI or placebo in children with a chronic cough.
  Arms: Sugar Pill

SUMMARY:
Cough is both an important physiologic component of lung defense and a cardinal indicator of disease. For those with chronic cough, defined as cough lasting for more than 3 weeks, the differential diagnosis is broad, including self-limited, persistent, and chronic diseases. The success of a given treatment depends upon a proper diagnosis, yet this is often not obvious. Gastroesophageal reflux (GER) has been proposed as one possible etiology of a chronic cough in a number of studies in the adult literature; nevertheless a clear cause and effect remains to be confirmed as there continues to be no gold standard test definitively to identify pathologic GER. Each year, billions of dollars are directed towards diagnosing and treating GER as it relates to adults and children with a chronic cough but without solid proof of effect.

We propose to test the null hypothesis that there is no causative role of GER with regards to the etiology of chronic cough in children. If the null hypothesis proves true, this has important medical and economic ramifications, as it would suggest that treatment of acid reflux for chronic cough in a child is unwarranted. With this conclusion, health care costs would be reduced and children spared inappropriate medication.

DETAILED DESCRIPTION:
Introduction

1.1. Cough

Cough is both an important physiologic component of lung defense and a cardinal indicator of disease. It is the second most common reason for medical visits during childhood. The metamorphosis of coughing from a normal to a pathologic event occurs along a gradient that includes frequency, character and duration.1 When considered with the age of the child, each of these characteristics informs decisions about diagnosis and management. For those with chronic cough, defined as cough lasting for more than 3 weeks2, the differential diagnosis is broad, including self-limited, persistent, and chronic diseases. An isolated cough in an otherwise healthy child may be secondary to recurrent viral bronchiolitis, post-infectious etiology, pertussis, cough variant asthma, post-nasal drip, or may be psychogenic in origin. Possible significant underlying causes of cough include cystic fibrosis, primary ciliary dyskinesia, immune deficiencies, chronic bronchitis, retained foreign bodies, airway lesions, tracheomalacia, or extrinsic compression of the airway3. Gastroesophageal reflux (GER) is also included in the differential diagnosis of chronic cough in children.

Specific Aims

1. To conduct a randomized , placebo controlled trial to test the null hypothesis that treatment of children with a chronic cough of more than 3 weeks' duration is not effected by medicine designed specifically to treat gastroesophageal reflux (GER) and its extraesophageal manifestations.
2. To utilize the "gold standard population"(identified through the protocol outlined in specific aim number 1) to use logistic regression analysis to identify which tests currently employed to identify GER can be employed within a statistically sound predictive model.

Patient Recruitment:

Children ages 2 to 18 years seen at the primary care pediatricians within one of the Massachusetts General Hospital for Children (MGHfC) associated practices with a chronic cough of three weeks or greater duration will be candidates for recruitment into the study. The MGHfC has approximately 260 community based pediatric practices within the greater Boston region. Children will also be recruited from the hospital based as well as satellite clinics of the divisions of Pediatric Gastroenterology and Pediatric Pulmonology at MGHfC as well as from the division of Pediatric Otolaryngology at the Massachusetts Eye and Ear Infirmary (MEEI).

Children will be evaluated first by their pediatricians and then by a team of Pediatric otolaryngologists, gastroenterologists, and pulmonologists for identifiable causes of their chronic cough. These children will be excluded from entry into proposed study. Children who 1) do not have an identifiable and treatable cause for their cough or 2) are suspected to have GER as a possible etiology of their cough as suggested by history and physical examination remain as candidates for recruitment.

Children in whom a clear diagnosis can not be established by the above described protocol then generally undergo a series of diagnostic endoscopies performed by the three clinical services simultaneously (as is current standard at the MEEI/MGHfC Pediatric Airway, Voice, and Swallowing Center) that include direct laryngoscopy, bronchoscopy with culture and bronchoalveolar lavage, esophagogastroduodenoscopy with biopsy, and placement of ambulatory impedance and double pH probe monitoring. It is at the this point when informed consent is taken for these procedures that the patients and their caregivers are recruited into the study at the Massachusetts Eye and Ear Infirmary. ( the site for the office and endoscopic visits). The point of randomization occurs at the time of endoscopy; administration of either PPI or placebo begins on the day following the endoscopy and continue for the three week time interval until the time of the first post-operative office visit.

Caregivers of children who are being scheduled for diagnostic endoscopy will be met by the P.I. (CJH) as well as by the nurse coordinator of the study who will review with them the Informed Consent Form and the Informed Assent Form for children over the age of 8 (as is standard at MEEI; informed consent forms will also be obtained from the caregivers of these children). A datasheet will be recorded for those caregivers who opt not to enter the study to identify why they did not enroll so these issues can potentially be addressed if there are issues with patient accrual and achieving adequate sample size.

Primary Study Objectives:

The primary study objectives are:

1. To compare the cough reduction rate using either PPI or placebo in children with a chronic cough
2. To compare the adverse events reported by the caregivers for their children who were treated with PPI therapy as opposed to placebo

The study design is based upon a non-parametric outcome variable and permits a Wilcoxon Rank Sum calculation. The proposed RCT is designed to provide 90% statistical power for showing a significant difference in clinical outcome attributable to PPI administration assuming a 5 point treatment difference on the summed questions from the CQ. The null hypothesis being tested is that there is no significant difference in the cough reduction rate between children with a chronic cough treated either with placebo or PPI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Children 2-18 years of age
2. Male and female children
3. Children of any race or ethnicity
4. Cough lasting longer than three weeks* * If a child has been placed on PPI or other antacid therapy for presumed but not documented extra-esophageal manifestations of GER, then these children will stop taking their antacid therapy after recruitment for the two-week interval between recruitment and the endoscopy, as is the standard protocol at MEEI to allow time for adequate "wash-out" prior to endoscopy and pH probe placement.

Exclusion Criteria:

1. The presence of a chronic respiratory, neurological or gastrointestinal disease and/or anomaly
2. An abnormal barium swallow study indicating vascular compression
3. Allergy with respiratory component,
4. Gross erosive esophagitis defined by EGD findings where patients will automatically be placed on PPI therapy without randomization

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
No primary outcome measure. | No timeframe.
  There is no primary outcome measure as this study was not activated. Therefore, no data was collected to measure or analyze.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary